CLINICAL TRIAL: NCT04554771
Title: Blood-borne Assessment of Stromal Activation in Esophageal Adenocarcinoma to Guide Tocilizumab Therapy: a Randomized Phase II Proof-of-concept Study
Brief Title: Blood-borne Assessment of Stromal Activation in Esophageal Adenocarcinoma to Guide Tocilizumab Therapy
Acronym: BASALT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Noordwest Ziekenhuisgroep (Other)
Responsible Party: Principal Investigator, Hanneke W. M. van Laarhoven, prof. dr. H.W.M. van Laarhoven, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL74310.018.20; 2020-002909-25 (EudraCT Number)
Record Dates: First submitted 2020-08-18; First posted 2020-09-18 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Esophageal Adenocarcinoma; Oesophageal Adenocarcinoma; Resectable Carcinoma
Keywords: Resectable; Esophageal adenocarcinoma; Neoadjuvant chemoradiation; Tocilizumab; Stroma activation
MeSH Terms: conditions — Adenocarcinoma Of Esophagus | interventions — tocilizumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Intervention Model Description: Randomized phase II proof-of-concept study with tocilizumab and standard of care paclitaxel, carboplatin and radiation followed by surgical resection of the oesophagus for patients with surgically resectable adenocarcinomas of the oesophagus or oesophageal junction. Patients will be grouped for serum ADAM12 with a cutoff of 203 ng/mL. Patients in both groups will be randomized to receive tocilizumab 8mg/kg on day 1, 15 and 29 or not in addition to paclitaxel 50mg/m2, carboplatin AUC 2 on day 1, 8, 15, 22 and 29 and radiation 41.4 Gy in 23 fractions. Surgery will be planned approximately in week 13-15, which is 8 to 10 weeks after the end of chemoradiation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ADAM12 high with tocilizumab and standard of care (Experimental): Patients have serum ADAM12 higher than 203ng/mL. Patients will receive tocilizumab 8 mg/kg with a maximum of 800 mg intravenously on day 1, 15 and 29 in addition to paclitaxel 50mg/m2 and carboplatin AUC 2 intravenously on day 1, 8, 15, 22 and 29. External beam radiation of 41.4 Gy will be given in 23 fractions. Surgery will be planned approximately in week 13-15, which is 8 to 10 weeks after the end of chemoradiation.
  Interventions: Drug: Tocilizumab 20 Mg/mL Intravenous Solution; Drug: Paclitaxel; Drug: Carboplatin; Radiation: External beam radiotherapy
- ADAM12 high with standard of care (Active Comparator): Patients have serum ADAM12 higher than 203ng/mL. Patients will receive paclitaxel 50mg/m2 and carboplatin AUC 2 intravenously on day 1, 8, 15, 22 and 29. External beam radiation of 41.4 Gy will be given in 23 fractions. Surgery will be planned approximately in week 13-15, which is 8 to 10 weeks after the end of chemoradiation.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Radiation: External beam radiotherapy
- ADAM12 low with tocilizumab and standard of care (Experimental): Patients have serum ADAM12 lower than 203ng/mL. Patients will receive tocilizumab 8 mg/kg with a maximum of 800 mg intravenously on day 1, 15 and 29 in addition to paclitaxel 50mg/m2 and carboplatin AUC 2 intravenously on day 1, 8, 15, 22 and 29. External beam radiation of 41.4 Gy will be given in 23 fractions. Surgery will be planned approximately in week 13-15, which is 8 to 10 weeks after the end of chemoradiation.
  Interventions: Drug: Tocilizumab 20 Mg/mL Intravenous Solution; Drug: Paclitaxel; Drug: Carboplatin; Radiation: External beam radiotherapy
- ADAM12 low with standard of care (Active Comparator): Patients have serum ADAM12 lower than 203ng/mL. Patients will receive paclitaxel 50mg/m2 and carboplatin AUC 2 intravenously on day 1, 8, 15, 22 and 29. External beam radiation of 41.4 Gy will be given in 23 fractions. Surgery will be planned approximately in week 13-15, which is 8 to 10 weeks after the end of chemoradiation.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Radiation: External beam radiotherapy

INTERVENTIONS:
Drug: Tocilizumab 20 Mg/mL Intravenous Solution — tocilizumab 8 mg/kg with a maximum of 800 mg intravenously on day 1, 15 and 29 of standard of care neoadjuvant chemoradiation
  Other Names: RoActemra; L04AC07
  Arms: ADAM12 high with tocilizumab and standard of care; ADAM12 low with tocilizumab and standard of care
Drug: Paclitaxel — Paclitaxel 50 mg/m2 will be given intravenously on days 1, 8, 15, 22 and 29
  Other Names: L01CD01
Drug: Carboplatin — Carboplatin AUC = 2 will be given intravenously on days 1, 8, 15, 22 and 29
  Other Names: L01XA02
Radiation: External beam radiotherapy — External beam radiotherapy will be delivered to a total dose of 41.4 Gy in 23 fractions of 1.8 Gy, 5 fractions per week starting the first day of the first cycle of chemotherapy

SUMMARY:
The primary objective of this study is to demonstrate that stroma-targeting by tocilizumab in patients with adenocarcinoma of the esophagus or gastroesophageal junction with highly activated stroma increases efficacy of chemoradiotherapy measured by pathological response according to the Mandard criteria. Patients will be grouped for ADAM12, a non-invasive blood-borne marker of stromal activation.

DETAILED DESCRIPTION:
Randomized phase II proof-of-concept study with tocilizumab and standard of care paclitaxel, carboplatin and radiation followed by surgical resection of the oesophagus for patients with surgically resectable adenocarcinomas of the oesophagus or oesophageal junction. Patients will be grouped for serum ADAM12 with a cutoff of 203 ng/mL. Patients in both groups will be randomized to receive tocilizumab 8mg/kg on day 1, 15 and 29 or not in addition to paclitaxel 50mg/m2, carboplatin dosed with area under the curve (AUC) 2 on day 1, 8, 15, 22 and 29 and radiation 41.4 Gy in 23 fractions. Surgery will be planned approximately in week 13-15, which is 8 to 10 weeks after the end of chemoradiation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma of the esophagus or gastroesophageal junction.
* Surgical resectable (<T4b, N0 or N+, M0), as determined by Endoscopic UltraSound (EUS) and/or CT scan of neck, thorax and abdomen. Tumors that cannot be passed with an endoscope for endoscopic ultrasound are eligible if all other criteria are fulfilled.
* T1N+ tumors are eligible.
* Tumor length longitudinal ≤ 10 cm; if larger than 10 cm, inclusion should be discussed with the principal investigator.
* If the tumor extends below the gastroesophageal (GE) junction into the proximal stomach, the bulk of the tumor must involve the esophagus or GE junction.
* Age ≥ 18.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Adequate hematological, renal and hepatic functions defined as:

  * neutrophiles ≥ 1.5 x 109/L
  * platelets ≥ 100 x 109/L
  * hemoglobin ≥ 5.6 mmol
  * total bilirubin ≤ 1.5 x upper normal limit
  * creatinine clearance (Cockroft) > 60 ml/min
* Written, voluntary informed consent
* Patients must be accessible to follow up and management in the treatment center

Exclusion Criteria:

* Past (within 5 years) or current history of malignancy other than entry diagnosis interfering with prognosis of esophageal cancer, not including superficial and adequately treated skin and cervical malignancies.
* Previous chemotherapy, radiotherapy and/or treatment with Interleukin-6 (IL6) receptor blockers for esophageal cancer
* Previous radiation to the mediastinum precluding full dose radiation of the currently present esophageal tumor.
* Previous chemotherapy and/or treatment with targeted agents and/or IL6 receptor blockers for other forms of cancer within the last six months.
* Invasion of the tracheobronchial tree or presence of tracheoesophageal fistula.
* T1N0 tumors or in situ carcinoma.
* Pregnancy (positive serum pregnancy test), planning to become pregnant, and lactation.
* Patient (male or female) is not willing to use highly effective methods of contraception (per institutional standard) during treatment and for 6 months (male or female) after the end of treatment.
* Clinically significant cardiovascular disease (including myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) precluding major surgery.
* Pulmonary fibrosis and/or severely impaired lung function precluding major surgery.
* Serious underlying medical condition which would impair the ability of the patient to receive the planned treatment, including prior allergic reactions to drugs containing Cremophor, such as teniposide or cyclosporine.
* Dementia or altered mental status that would prohibit the understanding and giving of informed consent
* Inadequate caloric- and/or fluid intake despite consultation of a dietician and/or tube feeding.
* Requires systemic treatment with IL6 receptor blockers or IL-6 antagonists, Tumor Necrosis Factor (TNF)-alpha blockers or other biologicals within the last six months before the first dose of trial treatment.
* Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy which has not resolved 3 days (simple infection such as cystitis) to 7 days (severe infection such as pyelonephritis) prior to the first dose of trial treatment.
* Has a total cholesterol > 6.5 mmol/L despite adequate treatment with lipid-lowering agents.
* Has evidence of (latent) tuberculosis infection in patient history.
* Receiving a live or live weakened vaccine during treatment with tocilizumab
* Has evidence of acute or chronic infection with hepatitis B
* Patients with prior allogeneic stem cell or solid organ transplantation.
* Pre-existing motor or sensory neurotoxicity greater than World Health Organization (WHO) grade 1.
* Known allergy for tocilizumab or one of its excipients (sucrose, polysorbate 80, disodium phosphate dodecahydrate, sodium dihydrogen phosphate dehydrate)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2028-04-10 (Estimated)

PRIMARY OUTCOMES:
Efficacy defined as pathological response to chemoradiotherapy according to the Mandard criteria | 34 months
  The primary outcome is efficacy of tocilizumab in patients with high and low stroma activation defined as pathological response according to the Mandard criteria

SECONDARY OUTCOMES:
R0 resection rate | 34 months
  Percentage of R0 resection at surgery
Progression free survival | 34 months
  Average time to progression of disease
Overall survival | 34 months
  average time to date of death
Interleukin 6- Signal Transducer and Activator of Transcription 3 (IL6-STAT3) pathway inhibition measured by gene expression analysis | 36 months
  Analysis of gene expression to measure level of inhibition of IL6-STAT3 pathway
IL6-STAT3 pathway inhibition measured by immunohistochemistry | 36 months
  Phosphorylated STAT3 and stromal abundance measured by immunohistochemistry in formalin-fixed paraffin-embedded tumor tissue
Levels of ADAM12 in tumor biopsies and serum | 36 months
  average levels of ADAM12 in tumor biopsies and serum
Incidence and severity of toxicity | 34 months
  Incidence of treatment-emergent adverse events according to CTCAE v5.0
Incidence and severity of radiation toxicity | 34 months
  Incidence of treatment-emergent adverse events according to Radiation Oncology Group (RTOG) criteria
Incidence and severity of post-operative complications | 36 months
  Incidence and severity of post-operative complications according to the Clavien - Dindo classification
Feasibility completion | 34 months
  Percentage completion of chemotherapy and radiation treatment
Feasibility withdrawal rate | 34 months
  Percentage withdrawal rate from surgery due to tocilizumab related complications
Feasibility delay | 36 months
  Percentage delay of surgery due to tocilizumab related complications

OTHER OUTCOMES:
Predictive biomarkers using oa RNA sequencing | 54 months
  Exploratory objectives are to identify additional predictive biomarkers based on tumor, fecal and blood samples. Among others we will use RNA sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Hanneke WM van Laarhoven, MD, PhD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Medical Oncology, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No